CLINICAL TRIAL: NCT03655509
Title: Searching a Dysfunction of Corticotropic and Thyrotropin Axis During the Acute Phase ( ≤48h ) of a Subarachnoid Hemorrhage Secondary to Spontaneous Rupture of Cerebral Aneurysm: Impact on the Incidence of Complications and Recovery at 1 Month
Brief Title: Searching a Dysfunction of Corticotropic & Thyrotropin Axis During the Acute Phase of a Subarachnoid Hemorrhage Secondary to Spontaneous Rupture of Cerebral Aneurysm
Acronym: HSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A01386-37
Record Dates: First submitted 2016-09-13; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-02

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACTH stimulation test (Other)
  Interventions: Procedure: Dynamic test ACTH stimulation

INTERVENTIONS:
Procedure: Dynamic test ACTH stimulation

SUMMARY:
Searching a dysfunction of corticotropic and thyrotropin axis during the acute phase ( ≤48h ) of a subarachnoid hemorrhage secondary to spontaneous rupture of cerebral aneurysm. Impact on the incidence of complications and recovery are evaluated at 1 month.

Blood sample are made within 48 hours of the onset of bleeding with assay of total plasma cortisol, plasma ACTH at 8 am and thyroid hormones (T3, free T4 , and TSH). Dynamic test ACTH stimulation (test Synacthene) with renewal of serum cortisol to H + 1 (60min). Evaluation in the first 30 days of the incidence of rebleeding, hydrocephalus, of vasospasm, infection and epilepsy. GOS to 1 month.

DETAILED DESCRIPTION:
Searching a dysfunction of corticotropic and thyrotropin axis during the acute phase ( ≤48h ) of a subarachnoid hemorrhage secondary to spontaneous rupture of cerebral aneurysm. Impact on the incidence of complications and recovery are evaluated at 1 month.

Blood sample are made within 48 hours of the onset of bleeding with assay of total plasma cortisol, plasma ACTH at 8 am and thyroid hormones (T3, free T4 , and TSH). Dynamic test ACTH stimulation (test Synacthene) with renewal of serum cortisol to H + 1 (60min). Evaluation in the first 30 days of the incidence of rebleeding, hydrocephalus, of vasospasm, infection and epilepsy. GOS to 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Acute phase ( ≤48h) of a subarachnoid hemorrhage secondary to spontaneous rupture of cerebral aneurysm (Glasgow coma scale >=9)

Exclusion Criteria:

* Pituitary failure
* Patient with corticosteroids drugs or antithyroid drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
ACTH stimulation test | 2 days
  ACTH stimulation test compared of threshold values at 48h

SECONDARY OUTCOMES:
ATCH levels | 2 days
  ATCH levels at 8 AM compared of threshold values at 48h
plasma cortisol | 2 days
  µg per L

IPD SHARING:
Plan to Share IPD: No